CLINICAL TRIAL: NCT00655486
Title: A Multicenter, Open-label Extension Trial to Assess the Long-term Safety and Tolerability of Lacosamide as Adjunctive Therapy in Subjects With Partial-onset Seizures
Brief Title: Study to Assess the Long-term Safety of Oral Lacosamide in Subjects With Partial-onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SP0926; 2014-004384-21 (EudraCT Number)
Expanded Access: NCT03559673 (No longer available)
Record Dates: First submitted 2008-03-26; First posted 2008-04-10 (Estimated); Results first posted 2011-07-15 (Estimated); Last update posted 2018-07-17 (Actual); Status verified 2017-07

CONDITIONS: Partial Epilepsies; Partial Onset Seizures
Keywords: Epilepsy; seizures; antiepileptic; Lacosamide; Vimpat; safety; adjunctive
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy; Seizures | interventions — Lacosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lacosamide (Experimental): Lacosamide 100 to 800 mg/day, flexible dosing, administered twice daily throughout the duration of the study (up to 2 years)
  Interventions: Drug: lacosamide

INTERVENTIONS:
Drug: lacosamide — Subjects' dose of lacosamide may be increased or decreased as needed to maintain a subject's effective and tolerable dose during the study. Tablets are 50 mg or 100 mg each; Dose is 100 mg/day up to 800 mg/day administered twice daily throughout the study (up to 2 years).
  Other Names: Vimpat

SUMMARY:
The purpose of this study is to allow eligible subjects from the parent study, SP925 [NCT00655551] to continue lacosamide and to obtain additional long-term safety data

DETAILED DESCRIPTION:
A multicenter, open-label extension study to assess the long-term safety and tolerability of lacosamide as adjunctive therapy in subjects with partial-onset seizures who were previously enrolled in the SP925 study [NCT00655551] (intravenous lacosamide loading dose followed by approximately 1 week of oral lacosamide maintenance).

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects who participated in SP925 [NCT00655551] for treatment of partial-onset seizures

Exclusion Criteria:

* Receiving any study drug or experimental device other than lacosamide
* Meets withdrawal criteria for parent study SP925 [NCT00655551]
* Experiencing ongoing serious adverse event

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 97 (Actual)
Dates: Start 2008-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (7):
- United States (7):
  - Phoenix, Arizona
  - Baltimore, Maryland
  - Chesterfield, Missouri
  - Columbus, Ohio
  - Philadelphia, Pennsylvania
  - Dallas, Texas
  - Charlottesville, Virginia

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started in April 2008 with enrollment occuring in the United States only. The study completed June 2010
Period: Overall Study
Arm/Group | Lacosamide
Started | 97
Completed | 69
Not Completed | 28
Not completed — Adverse Event | 10
Not completed — Lack of Efficacy | 8
Not completed — Withdrawal by Subject | 4
Not completed — Protocol Violation | 1
Not completed — Unsatisfactory compliance | 2
Not completed — Other: Pregnancy | 1
Not completed — Other: Could not tolerate BID dosing | 1
Not completed — Other: Abnormal electrocardiogram (ECG) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lacosamide
Number analyzed (Participants) | 97
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 95
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (11.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 50
Region of Enrollment [Number; unit: participants]
  United States | 97

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Adverse Event During This Open-label Extension Study (Maximum Study Duration 2 Years)
Description: An Adverse Event (AE) is any untoward medical occurrence (eg, noxious or pathological changes) in a subject or clinical investigation subject compared with pre-existing conditions, that occurs during any period of a clinical trial including Pre-treatment, Run-In, Wash-Out, or Follow-Up Periods. An AE is defined as being independent of assumption of any causality (eg, to study or concomitant medication, primary or concomitant disease, or study design).
Time Frame: 2 years
Population: All 97 subjects enrolled are in the Safety Set (SS) and are included in this analysis
Measure: Number; unit: subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 97
subjects | 93

2. Primary Outcome: Number of Subjects Who Withdrew From the Study Due to an Adverse Event (Maximum Study Duration 2 Years)
Description: as for outcome 1
Time Frame: 2 years
Population: All 97 subjects enrolled are in the Safety Set (SS) and are included in this analysis
Measure: Number; unit: subjects
Arm/Group | Lacosamide
Number analyzed (Participants) | 97
subjects | 10

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Lacosamide
Serious Adverse Events (participants affected / at risk) | 10/97
Other Adverse Events (participants affected / at risk) | 88/97
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=97)
Arrhythmia supraventricular (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Drug interaction (General disorders) | 1 (1)
Giardiasis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Post procedural bile leak (Injury, poisoning and procedural complications) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2)
Lethargy (Nervous system disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Homicidal ideation (Psychiatric disorders) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1)
Depression suicidal (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=97)
Tinnitus (Ear and labyrinth disorders) | 5 (5)
Diplopia (Eye disorders) | 17 (18)
Vision blurred (Eye disorders) | 10 (10)
Vomiting (Gastrointestinal disorders) | 16 (18)
Nausea (Gastrointestinal disorders) | 13 (14)
Diarrhoea (Gastrointestinal disorders) | 12 (13)
Constipation (Gastrointestinal disorders) | 5 (6)
Fatigue (General disorders) | 12 (12)
Chest pain (General disorders) | 8 (9)
Irritability (General disorders) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 14 (17)
Sinusitis (Infections and infestations) | 8 (11)
Urinary tract infection (Infections and infestations) | 7 (8)
Nasopharyngitis (Infections and infestations) | 6 (7)
Contusion (Injury, poisoning and procedural complications) | 5 (5)
Weight increased (Investigations) | 6 (6)
Dizziness (Nervous system disorders) | 43 (50)
Somnolence (Nervous system disorders) | 12 (13)
Coordination abnormal (Nervous system disorders) | 11 (13)
Headache (Nervous system disorders) | 11 (11)
Balance disorder (Nervous system disorders) | 11 (13)
Tremor (Nervous system disorders) | 8 (10)
Memory impairment (Nervous system disorders) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 5 (7)
Insomnia (Psychiatric disorders) | 9 (9)
Confusional state (Psychiatric disorders) | 8 (8)
Depression (Psychiatric disorders) | 7 (7)
Rash (Skin and subcutaneous tissue disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that is confidential and compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.